CLINICAL TRIAL: NCT00878787
Title: Theta-burst Transcranial Magnetic Stimulation for the Treatment of Childhood Dystonia and Spasticity
Brief Title: Theta-burst Transcranial Magnetic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Terence Sanger, Associate Professor, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SU-03162009-1999
Record Dates: First submitted 2009-03-20; First posted 2009-04-09 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Dystonia
MeSH Terms: conditions — Dystonia | interventions — Transcranial Magnetic Stimulation

ARMS (1):
- Theta-burst Trancranial Magnetic Stim (Experimental)
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation

SUMMARY:
Theta-burst transcranial magnetic stimulation (TBS) is a type of repetitive transcranial magnetic stimulation (rTMS) method that reduces the excitability of a small region of brain for less than one hour. Since dystonia and spasticity may be associated with increased excitability of motor cortex, we expect that by reducing the excitability of motor cortex with TBS we will temporarily improve these symptoms and hopefully open avenues in the future for the use of TBS as a new, non-invasive therapeutic intervention to aid in physical therapy and symptom amelioration of dystonia and spasticity. We will test for motor improvement during the hour immediately following TBS using tests of muscle function and quality of limb movement.

DETAILED DESCRIPTION:
Testing will occur at three identical visits, with escalating stimulation intensity at each visit. Initial screening will be performed by telephone or in clinic and final screening will be performed and informed consent will be signed at the start of the first study visit. Initial set-up and calibration of the magnetic stimulation device will require 10-20 minutes. Theta-burst stimulation requires 40 seconds. Hand and arm function will be tested immediately before and during the one hour following the TBS. Therefore, each visit should occupy 90-120 minutes. Each visit will be at least 2 days after the previous visit and a telephone call will be placed one week after the third visit.

Testing of limb function will be performed according to standard clinical rating scales, including the modified Ashworth spasticity scale and the Barry-Albright Dystonia rating scale. Electrophysiological testing of hand function will involve moving finger muscles against resistance while surface electromyographic signals (EMG) are monitored for the ability to activate one finger at a time while minimizing muscle co-contraction and overflow. Testing of arm function will involve measurement of the ability to relax the biceps and triceps and the resistance of the elbow to passive movement by the examiner.

Testing of cortical function will occur both before and after theta-burst stimulation, and will involve a standard protocol using suprathreshold single and paired-pulse magnetic stimulation with measurement of the induced motor evoked potential (MEP) in the hand and arm muscles. The resting MEP threshold and input-output curve will be measured for the first dorsal interosseus muscle. Paired-pulse inhibition of the MEP will be tested using a subthreshold pulse (80% of resting motor threshold) followed by a suprathreshold pulse at 2.5msec interval. Paired-pulse facilitation will be tested using a 12msec interval. Silent period duration in response to a pulse at 120% of resting motor threshold will be measured.

Theta-burst stimulation will be performed according to the standard protocols developed by Rothwell and co-workers with NIH and European consortium safety guidelines stringently enforced. Active motor threshold and resting motor threshold will be determined by single-pulse stimulation while monitoring electromyographic (EMG) activity at the first dorsal interosseus (FDI) muscle according to standard published protocols using commercially available surface EMG electrodes (DelSys Inc.). Stimulation will be performed using the commercially-available Magstim Rapid 2 (Magstim, Inc., Wales UK) with a standard figure-eight coil held by a member of the research team. Biphasic stimulation pulses will be given according to the standard included driver software. Single pulse, paired pulse, and theta-burst rapid stimulation protocols are directly available through standard user options on this device.

Threshold determination and stimulation location will be performed using each subject's most affected hand, or the non-dominant hand if both hands are affected. The location of lowest threshold for stimulation of the FDI will be determined by gradual movement of the stimulation coil over the surface of the contralateral scalp, in the region of the standard "C3" or "C4" electrode position (determined by international 10-20 EEG electrode placement convention). The handle of the stimulation coil will be pointed backward and 45 degrees from the sagittal plane so as to be approximately perpendicular to the rolandic fissure. The location of minimum threshold will be marked with a washable non-permanent marker on the subject's scalp in order to ensure consistency of stimulation.

For assessment of active motor threshold, subjects will be asked to contract the FDI muscle against resistance while being given biofeedback to maintain average integrated EMG at 20% of maximal voluntary isometric EMG. For assessment of resting motor threshold, EMG of the FDI must be less than 5% of maximal prior to stimulation. Single-pulses at increasing intensity will be used to determine the intensity at which 5 out of 10 pulses evoke an EMG response greater than 200mV (active threshold) or 50mV (resting threshold) above baseline. (Active motor threshold is virtually always less than the resting motor threshold. If this is not the case in a subject, then stimulation will be adjusted so that intensity never exceeds 80% of the resting motor threshold.) Thresholds will be assessed both before and after theta-burst stimulation, and these thresholds will be used for the cortical excitability testing as described above.

Stimulation intensity for theta burst will be set at 60% active motor threshold (visit 1), 80% active motor threshold (visit 2), and 80% resting motor threshold (visit 3). All stimulation is subthreshold, and thus not expected to produce muscle activity. To ensure this is the case, muscle activity will be continuously monitored from the FDI and stimulation will be aborted if any muscle activity during the TBS is detected.

Set-up of theta-burst stimulation will involve the same Magstim Rapid 2 device in which the handle of the stimulation coil (same standard figure-eight coil) will be pointed backward and 45 degrees from the sagittal plane so as to be approximately perpendicular to the rolandic fissure. We will use a continuous (cTBS) pattern of delivery for magnetic stimulation and pulses will occur in sets of three at 20msec intervals (50hz burst rate), with each burst of three pulses separated by 200msec (5hz inter-burst rate). Thus there are 15 pulses per second, divided into 5 bursts of three pulses. Each burst of three pulses will be the same. Stimulation will continue for 40 seconds, for a total of 600 pulses. The subject will be instructed to maintain all muscles relaxed, and relaxation relevant to stimulation will be monitored using EMG of the FDI muscle. After the initial TBS treatment, single and paired-pulse magnetic stimulation will be performed again to test cortical function and MEP threshold. These pulses will be applied in the same manner as before TBS treatment (described in previous paragraph).

The stimulation pulses can produce a loud clicking noise, and subjects will be provided with earplugs or sound isolating ear cuffs if the sound intensity becomes uncomfortable or exceeds normal speech volume.

ELIGIBILITY:
Inclusion Criteria:1. Dystonia affecting one or both hands or arms, and/or spasticity affecting one or both hands/arms 2. Age 2 years to 29 years 3. Sufficient cognitive function to attempt isolated finger movements Exclusion Criteria:1. any metallic implants in the head or neck 2. seizure within 2 years of study entry, or prior history of status epilepticus outside the newborn period.

3. deep-brain stimulator, vagal nerve stimulator, pacemaker, intrathecal baclofen pump, or other implanted electrical device.

4. prior neurosurgical procedure 5. migraine disorder 6. known cardiac arrhythmia, or history of syncope 7. use of tricyclic antidepressants or neuroleptic medications during the study 8. use or requirement for medications to treat seizures

Ages: 2 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
surface EMG overflow and control | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Terence D. Sanger, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States